CLINICAL TRIAL: NCT05228314
Title: A Phase 1, Observer-blind, Randomized, Controlled, Dose-finding Study to Evaluate the Safety and Immunogenicity of Clover Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2020S) in Adults 18 to 75 Years of Age
Brief Title: Safety and Immunogenicity Dose-finding Study of Adjuvanted SCB-2020S Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-2020S-002
Record Dates: First submitted 2021-12-24; First posted 2022-02-08 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCB-2019 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Standard dose SCB-2020S with CpG/alum adjuvant (Experimental): Day 1 and 22 standard dose of SCB-2020S with CpG/alum adjuvant
  Interventions: Biological: Candidate vaccine, SCB-2020S; Other: CpG/alum adjuvant
- Low dose SCB-2020S with low dose squalene based adjuvant (Experimental): Day 1 and 22 low dose of SCB-2020S with low dose squalene based adjuvant
  Interventions: Biological: Candidate vaccine, SCB-2020S; Other: Squalene based adjuvant
- Low dose SCB-2020S with standard dose squalene based adjuvant (Experimental): Day 1 and 22 low dose of SCB-2020S with standard dose squalene based adjuvant
  Interventions: Biological: Candidate vaccine, SCB-2020S; Other: Squalene based adjuvant
- Standard dose SCB-2020S with low dose squalene based adjuvant (Experimental): Day 1 and 22 standard dose of SCB-2020S with low dose squalene based adjuvant
  Interventions: Biological: Candidate vaccine, SCB-2020S; Other: Squalene based adjuvant
- Standard dose SCB-2020S with standard dose squalene based adjuvant (Experimental): Day 1 and 22 standard dose of SCB-2020S with standard dose squalene based adjuvant
  Interventions: Biological: Candidate vaccine, SCB-2020S; Other: Squalene based adjuvant
- Standard dose SCB-2019 with CpG/alum adjuvant (Active Comparator): Day 1 and 22 standard dose of SCB-20219 with standard CpG/alum adjuvant
  Interventions: Biological: Candidate vaccine, SCB-2019; Other: CpG/alum adjuvant

INTERVENTIONS:
Biological: Candidate vaccine, SCB-2020S — a recombinant SARS-CoV-2 trimeric S-protein (from beta variant) subunit vaccine for COVID-19
  Arms: Low dose SCB-2020S with low dose squalene based adjuvant; Low dose SCB-2020S with standard dose squalene based adjuvant; Standard dose SCB-2020S with CpG/alum adjuvant; Standard dose SCB-2020S with low dose squalene based adjuvant; Standard dose SCB-2020S with standard dose squalene based adjuvant
Biological: Candidate vaccine, SCB-2019 — a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19
  Arms: Standard dose SCB-2019 with CpG/alum adjuvant
Other: Squalene based adjuvant — Squalene based adjuvant
  Arms: Low dose SCB-2020S with low dose squalene based adjuvant; Low dose SCB-2020S with standard dose squalene based adjuvant; Standard dose SCB-2020S with low dose squalene based adjuvant; Standard dose SCB-2020S with standard dose squalene based adjuvant
Other: CpG/alum adjuvant — CpG/alum adjuvant
  Arms: Standard dose SCB-2019 with CpG/alum adjuvant; Standard dose SCB-2020S with CpG/alum adjuvant

SUMMARY:
This is a phase 1 study to assess the safety and immunogenicity of different formulations of the investigational adjuvanted recombinant SARS-CoV-2 trimeric S-protein (from beta variant) subunit vaccine (SCB-2020S vaccine), when administered as 2 dose vaccination series 21 days apart to adults ≥18 to ≤75 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 75 years of age
* Individuals are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests and other study procedures
* Individuals are willing and able to give an informed consent, prior to screening
* Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition.
* Female participants of childbearing potential may be enrolled in the study, if the participant has practiced highly effective method of contraception for 30 days prior to vaccination and has a negative pregnancy test on the day of vaccination and has agreed to continue adequate contraception for 3 months after the last vaccination
* Male participants must agree to employ acceptable contraception from the day of the first dose of the study vaccine until 6 months after the last dose of the study vaccine and also refrain from donating sperm during this period

Exclusion Criteria:

* Individuals with body temperature >37.8°C (axillary), or any acute illness at baseline (Day 1) or within 3 days prior to randomization.
* Body mass index at screening >30 kg/m2
* Individuals with laboratory-confirmed SARS-CoV-2 infection [as defined by reverse transcriptase polymerase chain reaction (RT-PCR) assay or Rapid COVID Antigen Test or an equivalent] at the screening visit or with known history of COVID-19 within 6 months prior to Day 1
* Individuals who have received an investigational or authorized COVID-19 vaccine within 6 months prior to Day 1, or plan to receive COVID-19 vaccine during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease [e.g., malignancy, human immunodeficiency virus (HIV) infection] or immunosuppressive/cytotoxic therapy (e.g., systemic corticosteroids, medications used for cancer chemotherapy, organ transplantation or to treat autoimmune disorders) within 3 months prior to Day 1.
* Individuals with any progressive unstable or uncontrolled clinical conditions
* Individuals who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or during the study period
* Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction, e.g., anaphylaxis to any components of the study vaccines
* Individuals who have a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix which have been cured, or other malignancies with minimal risk of recurrence).
* Individuals who have received any other investigational product within 30 days prior to Day 1 or intend to participate in another clinical study at any time during the conduct of this study
* Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 28 days after the second vaccination
* Individuals with known bleeding disorder that would, in the opinion of the investigator, contraindicate i.m. injection
* Individuals who have received treatment with rituximab or any other anti-CD20 monoclonal antibodies within 9 months prior to Day 1 or planned during the study period
* Administration of intravenous immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the study period
* Individuals with positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at Screening
* Individuals with safety laboratory test results (hematology, biochemistry, and coagulation) with a toxicity score of Grade ≥2 at Screening.
* The participant has a reported or documented history of alcohol abuse or drug addiction (excluding nonprescription health supplements and herbal remedies) within 1 year before the planned day of dose administration
* The participant has a positive test result for drugs of abuse at Screening
* Individuals with any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional risk to the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with local and systemic adverse events (AEs) after vaccination with SCB-2020S vaccine. | 7 days after each dose
  Proportion of subjects with solicited local and systemic adverse events
Number of participants with unsolicited AEs after vacccination with SCB-2020S vaccine | Up to 28 days after the last vaccination
  Proportion of subjects with unsolicited adverse events
Number of participants with MAAEs, SAEs, AESIs and AEs leading to discontinuation from study. | Up to 1 year after the last vaccination
  Proportion of participants with any adverse events in this category.
Number of participants with abnormal results in hematology parameters (hemoglobin, platelet count, red blood cell count, total and differential white blood cell count). | up to Day 29
  Proportion of participants with abnormal results in hematology parameters.
Number of participants with abnormal results in biochemistry parameters (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, blood urea nitrogen, creatinine, total protein). | up to Day 29
  Proportion of participants with abnormal results in biochemistry parameters.
Number of participants with abnormal results in coagulation parameters (activated partial thromboplastin, prothrombin time). | up to Day 29
  Proportion of participants with abnormal results in coagulation parameters.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibody (nAb) | Day 1, 22, 36, 90, 205 and 389
Proportion of participants achieving seroconversion for SARS-CoV-2 nAb | Day 22, 36, 90, 205 and 389
Geometric Mean Fold Rise (GMFRs) of SARS-CoV-2 nAb | Day 22, 36, 90, 205 and 389
Proportion of participants with nAb above a certain threshold | Day 1, 22, 36, 90, 205 and 389
GMT of SCB-2019 Binding Antibody | Day 1, 22, 36, 90, 205 and 389
Proportion of participants achieving seroconversion for SCB-2019 binding antibody | Day 22, 36, 90, 205 and 389
  SCR is the percentage of participants with a ≥4-fold increase in titer from that at Day 1 (or from LLoQ if Day 1 titer <LLoQ).
GMFR of SCB-2019 binding antibody | Day 22, 36, 90, 205 and 389
SCB-2019 binding antibody above lower limit of quantification. | Day 1, 22, 36, 90, 205 and 389

CONTACTS AND LOCATIONS:
Locations (3):
- South Africa (3):
  - Josha Research, Bloemfontein
  - Global Clinical Trials (Pty) Ltd, Pretoria
  - Wits Vaccines and Infectious Diseases Analytics (VIDA) Research Unit, Soweto